CLINICAL TRIAL: NCT03396029
Title: A Randomized Trial of Tailored Written Lifestyle Feedback in Colorectal Cancer Screening
Brief Title: Tailored Written Lifestyle Feedback in Colorectal Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Paula Berstad, Researcher, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2011/1272
Record Dates: First submitted 2017-12-29; First posted 2018-01-10 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Lifestyle; Diet Habit; Smoking Cessation; Physical Activity; Alcohol Drinking; Body Weight
Keywords: Lifestyle intervention; Diet; Smoking cessation; Physical activity; Alcohol; Body mass index; colorectal cancer screening; sigmoidoscopy
MeSH Terms: conditions — Feeding Behavior; Smoking Cessation; Motor Activity; Alcohol Drinking; Body Weight

STUDY DESIGN:
Who Masked: Investigator
Masking Description: A computer programme designed by the research team IT developer carried out the randomization. The recruitment and the contact between the investigators and the participants was mailed. There was no face-to-face contact.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Individually tailored lifestyle feedback (Experimental): Written, standardized individually tailored lifestyle feedback based on participants responses to a lifestyle questionnaire, and a leaflet on healthy lifestyle mailed to the participant.
  Interventions: Behavioral: Individually tailored lifestyle feedback; Behavioral: Standard leaflet
- Standard leaflet (Experimental): A leaflet on healthy lifestyle mailed to the participant.
  Interventions: Behavioral: Standard leaflet
- Control (No Intervention): No contact with the participant.

INTERVENTIONS:
Behavioral: Individually tailored lifestyle feedback — The written, standardized individually tailored lifestyle feedback includes feedback on consumption of fruit, berries and vegetables and alcohol, physical activity, smoking and body mass index.
  Arms: Individually tailored lifestyle feedback
Behavioral: Standard leaflet — The leaflet is The Norwegian Cancer Society's one-page information brochure on healthy lifestyle behaviours for low cancer risk, including non-smoking, healthy body weight, physical activity, diet, moderate alcohol consumption, moderate sun exposure etc.
  Arms: Individually tailored lifestyle feedback; Standard leaflet

SUMMARY:
This randomized controlled trial aims to investigate the effect of an individually tailored lifestyle feedback letter and a leaflet on lifestyle in the context of sigmoidoscopy screening.

DETAILED DESCRIPTION:
Cancer screening may be used as a teachable moment for healthy lifestyle behaviours. This study aims to investigate the effect of minimal, but individually tailored lifestyle advice and a standard leaflet on healthy lifestyle given at a colorectal cancer screening context on one-year changes in these behaviours in a population-based sample of men and women.

Individuals invited to sigmoidoscopy screening in the piloting of Norwegian Bowel Cancer Screening are additionally invited to this lifestyle intervention study. Changes in lifestyle are measured by a brief lifestyle questionnaire administered at prescreening and after one year. The intervention to the intervention arms is given after completion of the prescreening lifestyle questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Invited to sigmoidoscopy screening in the Norwegian Bowel Cancer Screening Pilot Study

Exclusion Criteria:

* Excluded from sigmoidoscopy screening due to medical reasons, previous colorectal cancer diagnosis, relocating out of the screening municipalities or previous colonoscopy in the last 12 months.

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3642 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2016-10-30 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
A questionnaire-based lifestyle score | One year; from pre-screening until one year after
  A score variable ranging from 0 (least favorable) to 6 (most favorable), calculated as the sum of self-reported favorable lifestyle factors assessed by a questionnaire; non-smoking (1 score point), body mass index less than 25 kg/m2 (1 score point), a minimum of seven physical activity sessions of 30 minutes per a week (1 score point), a maximum of four dinner servings of red and processed meat per a week (1 score point), a minimum of three servings of fruit, berries and vegetables per a day (0.5 score point) and a minimum of one serving of fatty fish per a week (0.5 score points)

SECONDARY OUTCOMES:
Smoking status | One year; from pre-screening until one year after
  Self-reported smoking status (smoking vs. non-smoking), assessed by a questionnaire
Alcohol consumption | One year; from pre-screening until one year after
  Self-reported consumption of alcoholic beverages (glasses/week), assessed by a questionnaire
Physical activity | One year; from pre-screening until one year after
  Self-reported weekly time spent in physical activity (number of 30-minute activity sessions per week), assessed by a questionnaire
Consumption of fruit and vegetables | One year; from pre-screening until one year after
  Self-reported consumption of fruit, berries and vegetables (servings per day), assessed by a questionnaire
Body weight | One year; from pre-screening until one year after
  Self-reported body weight (whole kilograms), assessed by a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Paula Berstad, PhD, Principal Investigator — Norwegian Institute of Public Health

IPD SHARING:
Plan to Share IPD: No